CLINICAL TRIAL: NCT02083328
Title: Influence of Caffeine on Heart Rate Variability and Exercise Performance in in Tetraplegic and Paraplegic Subjects Compared to Able-bodied Subjects
Brief Title: Influence of Caffeine on HRV and Exercise Performance in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-03
Record Dates: First submitted 2014-03-06; First posted 2014-03-11 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Caffeine; Spinal Cord Injury
Keywords: heart rate variability; exercise performance
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Caffeine; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Active Comparator): Caffeine will be administrated at a dosage of 6mg/kg of body mass. It is ingested once, one hour before the exercise performance test.
  Interventions: Dietary Supplement: Caffeine
- Mannitol (Placebo) (Placebo Comparator): Placebo capsules will be administrated one hour before the exercise performance test. The subject gets exactly the same number of capsules as for the caffeine dosage. Caffeine and placebo capsules look the same.
  Interventions: Dietary Supplement: Placebo (Mannitol)

INTERVENTIONS:
Dietary Supplement: Caffeine — Caffeine will be filled in gelatine capsules and administrated in a dosage of 6mg per kg body mass
  Arms: Caffeine
Dietary Supplement: Placebo (Mannitol) — Mannitol filled in gelatine capsules
  Arms: Mannitol (Placebo)

SUMMARY:
The aim is to investigate the influence of caffeine on heart rate variability and on performance in a 3 min exercise test in different population groups (able-bodied, paraplegic and tetraplegic subjects).

In general, the investigators are interested in the differences between the heart rate variability before and after caffeine supplementation and if the subjects exercise performance is enhanced using this type of supplementation. Another objective is to see whether there are differences between able-bodied and disabled subjects.

Tetraplegic subjects showed in some previous studies no Low-Frequency-component (LF) for heart rate variability and no increase in catecholamines after the ingestion of caffeine. Therefore the investigators think, that tetraplegic subjects won't show any ergogenic effect in exercise performance after the intake of caffeine. On the other hand, paraplegic subjects should show similar differences of heart rate variability after the ingestion of caffeine as able-bodied subjects. Paraplegic subjects should benefit from caffeine supplementation in an increase in exercise performance.

DETAILED DESCRIPTION:
This study will be conducted in a placebo-controlled, double-blind and randomised study protocol. Every subject has to undergo three test session at the sports medicine in Nottwil. At the first visit, the investigators will check the subjects fitness using a health questionnaire with specific question about diseases and family health history. Additionally, subjects has to perform a maximal exercise test (ramp protocol at the arm crank ergometer) to measure maximal oxygen uptake, maximal heart rate and maximal power output. After a little break, subjects have to perform a familiarization trial at the arm crank ergometer. They have to perform exactly the same test as they have to perform later in the two test sessions.

Minimum two days later the subjects visits the sports medicine Nottwil for the first test session. At first, they have to answer some specific question about sleep, recent training, recent nutritional intake and the actual health condition. Afterwards, they have to lie down for a 10min rest where after 9min blood pressure will be measured. With a heart rate monitor HRV will be measured during 5 min in supine position and afterwards during 6 min in sitting position. Metronomic breathing (15x/min) is mandatory and will be simulated through a metronome. During the HRV measurement also tidal volume will be measured. As the first HRV measurement session is finished, a blood withdrawal will be taken to measure catecholamine concentrations. Then, when all these measurements are completed, a supplement (either caffeine or the placebo) will be ingested in gelatine capsules. After the ingestion of these capsules, the subject has a 40 min break where they can read something or just relax. During these 40 min physical activity or the ingestion of any nutrition is prohibited.

After these 40min, the second HRV measurement starts. The process of this measurement is exactly the same as for the first HRV measurement. They lay down for a 10min rest with blood pressure measurement after 9 min. Afterwards again a 5min HRV measurement in supine position and a 6min measurement in sitting position. Tidal volume is measured during this HRV measurement.

When this second HRV measurement session is finished, a second blood withdrawal has to be taken. That means, one hour after the ingestion of either placebo or caffeine, catecholamine are analysed for a second time. If the blood is taken, the warm up can start. After the standardised warm up lactate concentration of the blood is analysed taking 10 ul of blood from the earlobe. The subject will be asked to evaluate the warm up with the rate of perceived exertion (following the Borg scale). If everything is in order, the 3min exercise test can start. During this test, respiratory parameters will be measured using an Oxycon Pro device (device to measure oxygen consumption). Just after having finished these 3 min of exercising, for a second time lactate concentration will be measured and again they have to rate the exertion using the Borg scale.

After a short 5min break the third HRV measurement starts. Again HRV will be measured during a 5min time in supine position and a 6min time in sitting position. Tidal volume will be measured during the whole HRV measurement. With this HRV measurement the first test session is finished and a second test session will be conducted at least more than two days later in a randomised manner.

The first session with the familiarization trial will be finished in around 75 min. For the two test sessions the subject has to be at the sports medicine for around 2 hours.

In the following chart, the test sessions are visually displayed. The administrated dose of caffeine is defined to 6mg per kg bodyweight for all our subjects. Caffeine will be filled in gelatine capsules.

Also the placebo (Mannitol) will be filled in gelatine capsules and the subjects have to ingest the same amount of capsules for both supplements.

30 subjects will be tested in total. In each group 10 subjects will participate. That means 10 healthy able-bodied subjects, 10 tetraplegic (C5-7, American Impairment Score (AIS) A) and 10 paraplegic (sub Th8, AIS A) subjects will be tested. As it is not easy to find 10 physically active, completely injured tetraplegic subjects, a number of 10 subjects should be sufficient for this pilot study.

As the investigators know from previous studies conducted with disabled subjects, the level of the lesion is one critical point. Therefore, the investigators tried to include subjects with almost the same lesion level and all sensory and motoric completely lesioned. This could aid us to have more homogenous groups of different populations.

Inclusion criteria: healthy, non-smoking men, minimal 3x45min physical activity per week, tetraplegic (C5 to C7) or paraplegic (sub Th8), complete lesion, more than 6 month after rehabilitation program Exclusion: drugs or supplements which influences heart rate variability, Diabetes

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Age between 18 and 60 years
* Healthy, non-smoking men
* Tetraplegic subjects: C5-7, AIS A (sensory and motoric complete injury)
* Paraplegic subjects: sub Th8, AIS A (sensory and motoric complete injury)
* Min. 3x45min physical activity per week

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Caffeine 12 hours before the test session
* Women
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Diabetes
* Less than 7 hours of sleep in the nights before the exercise testing
* Not following the nutrition guidelines (no standardised nutrition)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Exercise performance | during 3min of arm cranking over a 2 week period
  An exercise performance test of 3min will be performed at an arm crank ergometer to measure exercise performance output after the ingestion of a placebo or caffeine supplement.

SECONDARY OUTCOMES:
Heart rate variability (HRV) before the ingestion of supplement | over 2 weeks
  HRV measurement is conducted before the ingestion of any supplement (caffeine or placebo)
Heart rate variability (HRV) after the exercise performance test | over 2 weeks of study phase
  HRV measurement is conducted 5min after the exercise performance test
Catecholamine | over 2 weeks
  A blood withdrawal is taken before the ingestion of any supplement to analyse epinephrine and norepinephrine concentration in the blood.
Heart rate variability 40min after the ingestion | 40min after the ingestion
  HRV will be measured 40min after the ingestion of the supplement

OTHER OUTCOMES:
Blood pressure | over 2 weeks of study phase
  Blood pressure measured before the ingestion of any supplement (caffeine or placebo)
Blood pressure | 40min after the ingestion of the supplement
  Blood pressure measured 40min after the ingestion of any supplement (caffeine or placebo)
Heart rate | during the 3min exercise test
  Heart rate will be measured during the 3min exercise performance test
Tidal volume | over 2 weeks of study phase
  Tidal volume will be measured during the HRV measurements
Rate of perceived exertion | after the 3min exercise performance test
  Rate of perceived exertion will be measured after the 3min exercise performance test using the Borg scale (6-20)
Lactate concentration | after the 3min exercise performance test
  Lactate concentration will be measured after the exercise performance test.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Perret, Dr. sc. nat., Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (1):
- Sports Medicine Nottwil, Nottwil, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Flueck JL, Schaufelberger F, Lienert M, Schafer Olstad D, Wilhelm M, Perret C. Acute Effects of Caffeine on Heart Rate Variability, Blood Pressure and Tidal Volume in Paraplegic and Tetraplegic Compared to Able-Bodied Individuals: A Randomized, Blinded Trial. PLoS One. 2016 Oct 24;11(10):e0165034. doi: 10.1371/journal.pone.0165034. eCollection 2016. PMID 27776149